CLINICAL TRIAL: NCT00004758
Title: Phase II Randomized Study of Early Surgery Vs Multiple Sequential Antiepileptic Drug Therapy for Infantile Spasms Refractory to Standard Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of California, Los Angeles (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/11691; UCLA-9508342
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Spasms, Infantile; Epilepsy
Keywords: infantile spasms; epilepsy; neurologic and psychiatric disorders; rare disease; seizures
MeSH Terms: conditions — Spasms, Infantile; Epilepsy; Neurologic Manifestations; Mental Disorders; Rare Diseases; Seizures | interventions — Carbamazepine; Adrenocorticotropic Hormone; Nitrazepam; Pyridoxine; Valproic Acid; Surgical Procedures, Operative

INTERVENTIONS:
Drug: carbamazepine
Drug: corticotropin
Drug: nitrazepam
Drug: pyridoxine
Drug: valproic acid
Procedure: Surgery

SUMMARY:
OBJECTIVES: I. Evaluate the efficacy of surgical resection of an identifiable zone of cortical abnormality versus multiple drug therapy in children with infantile spasms refractory to standard therapy.

II. Assess how infantile spasms interfere with development and whether this is partially reversible.

III. Determine the predictors of good surgical outcome and whether surgery permanently controls seizures and improves development.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients are randomly assigned to 1 of 2 treatment groups. The first group undergoes sequential antiepileptic therapy with pyridoxine, corticotropin, valproic acid, carbamazepine, and nitrazepam. The sequence of administration may be altered based on drugs taken prior to entry. Any drug may be omitted due to medical contraindications or prior use at study doses or higher.

The second group undergoes surgical resection of the zone of cortical abnormality. A functional hemispherectomy is performed for hemiparesis or diffuse unihemispheric dysfunction.

If seizures are controlled in the first group at 3 months, the current medication is maintained; if seizures are not controlled, sequential therapy continues to completion. Patients experiencing uncontrolled seizures at 6 months cross to surgery.

Surgical patients experiencing uncontrolled seizures at 3 months or persistent seizures after taper of pre-study antiepileptics cross to drug therapy.

All patients are followed at 6 months and 1, 2, 3, 5, 7, and 10 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Disease Characteristics

* Infantile spasms or seizures with diagnosis based on the following: short muscular contractions leading to flexion or extension; Single or repetitive electroencephalogram (EEG) consistent with diagnosis, i.e., hypsarrhythmia, modified hypsarrhythmia, multifocal spike and wave abnormalities; developmental quotient less than 70
* Zone of cortical abnormality in 1 lobe, contiguous multilobes, or 1 hemisphere; confirmed by historical, neurological, and physical evidence, including EEG, closed circuit televised EEG, computed tomography, magnetic resonance imaging, and/or positron-emission tomography; at least 2 abnormal test/imaging results required
* No treatable seizure etiology such as metabolic disease or infection

Prior/Concurrent Therapy

* Failed standard therapy, i.e., refractory to corticotropin (at least 40 IU/day for 14 days) as follows: persistent infantile spasms OR recurrent spasms after discontinuation or taper OR complications requiring dose modification
* At least 1 month of standard antiepileptic drug with documented therapeutic blood levels

Patient Characteristics

* No medical contraindication to surgery
* English-speaking family

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 1993-11

CONTACTS AND LOCATIONS:
Overall Officials: W. Donald Shields, Study Chair — University of California, Los Angeles